CLINICAL TRIAL: NCT00667459
Title: A Prospective, Multicenter, Controlled Clinical Trial of an Artificial Cervical Disc LP at a Single Level for Symptomatic Cervical Disc Disease
Brief Title: Study of Safety & Effectiveness of PRESTIGE® LP Cervical Disc vs. Anterior Cervical Fusion in Cervical DDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESTIGE® LP Protocol, #P03-03
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Cervical Degenerative Disc Disease
Keywords: Cervical Disc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational (Experimental): PRESTIGE® LP Cervical Disc
  Interventions: Device: PRESTIGE® LP Cervical Disc
- Control (Active Comparator): Control patients who received a ACDF fusion treatment from a previous IDE trial (NCT00642876)
  Interventions: Device: ATLANTIS Anterior Cervical Plate

INTERVENTIONS:
Device: PRESTIGE® LP Cervical Disc — The PRESTIGE® LP Cervical Disc was inserted into the intervertebral disc space of the cervical spine using the anterior surgical approach.
  Other Names: PRESTIGE® LP
  Arms: Investigational
Device: ATLANTIS Anterior Cervical Plate — Anterior cervical discectomy and fusion with ATLANTIS plate for control group
  Other Names: ATLANTIS plate
  Arms: Control

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and effectiveness of the PRESTIGE® LP Cervical Disc as a method of treating patients with symptoms of cervical degenerative disc disease at a single level from C3-C4 to C6-C7.

DETAILED DESCRIPTION:
This pivotal clinical trial was conducted to compare treatment data of the investigational implant device,the PRESTIGE® LP Cervical Disc, with a control patient group receiving a plate. The PRESTIGE® LP Cervical Disc devices were implanted using an anterior surgical approach. Data from control patients receiving anterior cervical discectomy and fusion with an ATLANTIS Anterior Cervical Plate from the initial Artificial Cervical Disc study (NCT00642876) were compared as both treatment groups receive single-level surgical treatment from C3-C4 to C6-C7 for symptomatic cervical degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

* Has cervical degenerative disc disease as defined as: intractable radiculopathy and/or myelopathy with at least one of the following items producing symptomatic nerve root and/or spinal cord compression that is documented by patient history: a) herniated disc; b) osteophyte formation
* One level requiring surgical treatment
* C3-C4 disc to C6-C7 disc level involvement
* Unresponsive to non-operative treatment for six weeks or presence of progressive symptoms or signs of cord compression
* No previous surgical procedures at the involved level or any planned surgical procedure at the involved or adjacent level.
* Preop Neck Disability index score ≥ 30
* Preop Neck Pain score of ≥ 20 based on the Preop Neck & Arm Pain Questionnaire
* Not pregnant at time of surgery
* Willing and able to comply with study plan and able to understand and sign patient informed consent

Exclusion Criteria:

* Any other cervical spinal condition requiring surgical treatment at the involved level
* Documented or diagnosed cervical instability defined by radiographs showing

  1. Sagittal plane translation > 3.5mm or
  2. Sagittal plane angulation > 20 degrees.
* More than one cervical level requiring surgery
* A fused level adjacent to the level to be treated
* Severe pathology of the facet joint of involved bodies
* Previous surgery at the involved level
* Previously diagnosed osteopenia or osteomalacia
* Any of the following that may be associated with an osteoporosis diagnosis (if "Yes" to any of these, a DEXA Scan will be required to determine eligibility)

  1. Postmenopausal non-Black female over 60 years of age and weighs less than 140 pounds
  2. Postmenopausal female that has sustained a non-traumatic hip, spine, or wrist fracture
  3. Male over the age of 70
  4. Male over the age of 60 that has sustained a non-traumatic hip or spine fracture.

If the level of Bone Mineral Density is a T score of -3.5 or lower or a T score of -2.5 or lower with the vertebral crush fracture, then the patient is excluded.

* Presence of spinal metastases
* Overt or active bacterial infection, either local or systemic
* Severe insulin dependent diabetes
* Chronic or acute renal failure or history of renal disease
* Temperature > 101º F oral at surgery
* Documented allergy to stainless steel, titanium or a titanium alloy
* Mentally incompetent
* Is a prisoner
* Is pregnant
* Is an alcohol and/or drug abuser
* Has received drugs which may interfere with bone metabolism within 2 weeks prior to the planned surgery date (steroids, methotrexate), excluding routine preop anti-inflammatories)
* A history of endocrine or metabolic disorder known to affect osteogenesis
* A condition that requires postop medications that interfere with the stability of the implant (steroids). This does not include low dose aspirin therapy.
* Received treatment with an investigational therapy within 28 days prior to surgery or planned for 16 weeks following implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Emory Orthopaedics and Spine Center, Atlanta, Georgia
  - The Hughston Clinic, P.C., Columbus, Georgia
  - Coeur d'Alene Spine and Brain, PLLC, Coeur d'Alene, Idaho
  - Central Illinois Neuroscience, Bloomington, Illinois
  - Indiana Spine, Carmel, Indiana
  - OrthoIndy, Indianapolis, Indiana
  - Cedar Neurological Surgeons, PC, Cedar Rapids, Iowa
  - Sports Medicine North, Peabody, Massachusetts
  - The Orthopaedic Center of St. Louis, Chesterfield, Missouri
  - Springfield Neurological Institute, Springfield, Missouri
  - Buffalo Neurosurgery Group, West Seneca, New York
  - NeuroSpine Institute, LLC, Eugene, Oregon
  - Clinical Trials for South Carolina, Charleston, South Carolina
  - Chattanooga Orthopaedic Group, Chattanooga, Tennessee
  - Brain and Spine Center of Texas, L.L.P., Plano, Texas
  - University of Virginia,Neurosurgery Department, Charlottesville, Virginia

REFERENCES:
- [Derived] Gornet MF, Lanman TH, Burkus JK, Hodges SD, McConnell JR, Dryer RF, Schranck FW, Copay AG. One-Level Versus 2-Level Treatment With Cervical Disc Arthroplasty or Fusion: Outcomes Up to 7 Years. Int J Spine Surg. 2019 Dec 31;13(6):551-560. doi: 10.14444/6076. eCollection 2019 Dec. PMID 31970051
- [Derived] Gornet MF, Burkus JK, Shaffrey ME, Schranck FW, Copay AG. Cervical disc arthroplasty: 10-year outcomes of the Prestige LP cervical disc at a single level. J Neurosurg Spine. 2019 May 10;31(3):317-325. doi: 10.3171/2019.2.SPINE1956. Print 2019 Sep 1. PMID 31075769
- [Derived] Gornet MF, Burkus JK, Shaffrey ME, Nian H, Harrell FE Jr. Cervical Disc Arthroplasty with Prestige LP Disc Versus Anterior Cervical Discectomy and Fusion: Seven-Year Outcomes. Int J Spine Surg. 2016 Jun 22;10:24. doi: 10.14444/3024. eCollection 2016. PMID 27441182

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Control patients who received ACDF fusion treatment from a previous IDE trial (NCT00642876)
Period: Overall Study
Arm/Group | Investigational | Control
Started | 280 | 265
Completed | 272 | 220
Not Completed | 8 | 45
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 8 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational | Control | Total
Number analyzed (Participants) | 280 | 265 | 545
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (8.8) | 43.9 (8.8) | 44.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 143 | 294
  Male | 129 | 122 | 251
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 271 | 243 | 514
  Black | 7 | 13 | 20
  Asian | 0 | 2 | 2
  Hispanic | 1 | 6 | 7
  Other | 1 | 1 | 2
Height [Mean (Standard Deviation); unit: in.] | 67.7 (4.1) | 67.5 (4.2) | 67.6 (4.2)
Weight [Mean (Standard Deviation); unit: lbs.] | 186.9 (45.0) | 184.7 (41.5) | 185.8 (43.3)
Marital Status [Number; unit: participants]
  Single | 40 | 32 | 72
  Married | 189 | 204 | 393
  Divorced | 42 | 24 | 66
  Separated | 7 | 3 | 10
  Widowed | 2 | 2 | 4
Education Level [Number; unit: participants]
  < High School | 15 | 14 | 29
  High School | 57 | 77 | 134
  > High School | 206 | 173 | 379
  Unknown | 2 | 1 | 3
Worker's Compensation Case [Number; unit: participants]
  Yes | 32 | 35 | 67
  No | 248 | 230 | 478
Unresolved Spinal Litigation [Number; unit: participants]
  Yes | 34 | 32 | 66
  No | 246 | 233 | 479
Tobacco Used [Number; unit: participants]
  Yes | 74 | 92 | 166
  No | 206 | 173 | 379
Alcohol Used [Number; unit: participants]
  Yes | 150 | 141 | 291
  No | 130 | 124 | 254
Preop Work Status [Number; unit: participants]
  Yes | 188 | 166 | 354
  No | 92 | 99 | 191

OUTCOME MEASURES:

1. Primary Outcome: Rate of Overall Success
Description: Rate of overall success is reported as the percentage of participants who met all of the following criteria:
  1. Postoperative Neck Disability Index score improvement of at least a 15-points from preoperative;
  2. Maintenance or improvement in neurological status;
  3. Disc height success which was defined as either the anterior or posterior measurements meeting the criteria of "Postoperative Height - 6 Week Postoperative Height ≥ -2mm";
  4. No serious adverse event classified as implant associated or implant/surgical procedure associated; and
  5. No secondary surgical procedure classified as a "failure."
Time Frame: 24 months
Population: The primary analysis dataset for this study consists of all subjects who received study devices and completed the initial surgical procedures. The analysis was based on the observed data and missing data due to lost-to-follow-ups were imputed. For the primary endpoint, the analysis consists of 226 investigational subjects and 171 control subjects.
Measure: Number; unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 226 | 171
percentage of participants | 70.4 | 63.2
Statistical Analysis 1: Comparison: Investigational vs Control; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the overall success rates in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P(p1 - p0 > -d | data) be at least 0.95, then the null noninferiority hypothesis will be rejected, and non-inferiority of the investigational device to the control will be claimed; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is 0.1; p = 0.995, Bayesian logistic model — The posterior probably of non-inferiority was calculated and presented instead of the p-value; The propensity score method was used to adjust possible effects on outcomes caused by differences in baseline characteristic due to non-randomization; Risk Difference (RD) = 0.032, 95% CI 2-sided [-0.070 to 0.134] — The posterior mean of P1-P0, along with the corresponding 95% highest posterior density (HPD) interval was presented instead of the usual 95% CI
Statistical Analysis 2: Comparison: Investigational vs Control; Superiority comparison of success rates in two treatment groups was a secondary objective of this trial. Superiority analysis was performed if non-inferiority was demonstrated. If the posterior probability is at least 0.95, a claim of superiority can be made; Test type: Superiority or Other; p = 0.736, Bayesian logistic model — The posterior probably of superiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Success Rate of Neck Disability Index
Description: Success rate of Neck Disability Index is reported as the percentage of participants whose neck disability index score met: Pre-treatment Score - Post-treatment Score ≥ 15.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable NDI success status at 24 months, which leads to 270 subjects in the investigational group and 219 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 270 | 219
percentage of participants | 87.8 | 80.8
Statistical Analysis 1: Comparison: Investigational vs Control; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the success rates of NDI in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P(p1 - p0 > -d | data) be at least 0.95, then the null noninferiority hypothesis will be rejected, and non-inferiority of the investigational group will be claimed for this endpoint; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 1.0, Bayesian logistic model — The posterior probably of non-inferiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 0.048, 95% CI 2-sided [-0.020 to 0.118] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Investigational vs Control; Superiority comparison of success rates in two treatment groups was a secondary objective of this trial. Superiority analysis was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.912, Bayesian logistic model — The posterior probably of superiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Success Rate of Neurological Status
Description: Success rate of neurological status is reported as the percentage of participants who met neurological success defined as maintenance or improvement in all sections (motor, sensory, and reflexes) for the time period evaluated. In order for a section to be considered a success, each element in the section must remain the same or improve from the time of the preoperative evaluation to the time period evaluated.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable neurological success status at 24 months, which leads to 270 subjects in the investigational group and 220 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 270 | 220
percentage of participants | 93.3 | 83.6
Statistical Analysis 1: Comparison: Investigational vs Control; The null hypothesis H0: p1 + d ≤ p0, and the alternative hypothesis is Ha: p1 + d > p0 where P0 and P1 are the overall success rates in the control group and the investigational group respectively, and d is the non-inferiority margin. The analyses used Bayesian methodology. Should the posterior probability P (p1 - p0 > -d | data) be at least 0.95, then the null non-inferiority hypothesis will be rejected, and non-inferiority of the investigational device to the control will be claimed; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 1.0, Bayesian logistic model — The posterior probably of non-inferiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 0.099, 95% CI 2-sided [0.038 to 0.161] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Investigational vs Control; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.999, Bayesian logistic model — The posterior probably of superiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Rate of Disc Height Success
Description: Disc height was assessed by determining the Functional Spinal Unit (FSU) height. The rate of disc height success is reported as the percentage of participants whose disc height for each level based on either the anterior or posterior measurements met the following criterion: Postoperative Height - 6 Week Postoperative Height >= -2mm
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable disc height success (FSU success) status at 24 months, which leads to 224 subjects in the investigational group and 164 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 224 | 164
percentage of participants | 91.5 | 95.1
Statistical Analysis 1: Comparison: Investigational vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 0.992, Bayesian logistic model — The posterior probably of non-inferiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -0.034, 95% CI 2-sided [-0.085 to 0.021] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Investigational vs Control; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.097, Bayesian logistic model — The posterior probably of superiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Neck Pain Success Rate
Description: Numerical rating scales were used to evaluate pain intensity and frequency. The pain score (0 min, 100 max) was derived by multiplying the numerical rating scores from the pain intensity (0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be.") and frequency scales (0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time"). Neck pain success rate is reported as the percentage of participants whose neck pain improvement met: Preoperative Score - Postoperative Score > 0.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable neck pain success status at 24 months, which leads to 270 subjects in the investigational group and 219 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 270 | 219
percentage of participants | 96.3 | 97.3
Statistical Analysis 1: Comparison: Investigational vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 1.0, Bayesian logistic model — The posterior probably of non-inferiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -0.010, 95% CI 2-sided [-0.043 to 0.023] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Investigational vs Control; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.273, Bayesian logistic model — The posterior probably of superiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Arm Pain Success Rate
Description: Numerical rating scales were used to evaluate pain intensity and frequency. The pain score (0 min, 100 max) was derived by multiplying the numerical rating scores from the pain intensity (0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be.") and frequency scales (0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time"). Arm pain success rate is reported as the percentage of participants whose arm pain improvement met: Preoperative Score - Postoperative Score > 0.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable arm pain success status at 24 months, which leads to 268 subjects in the investigational group and 219 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 268 | 219
percentage of participants | 96.3 | 95.0
Statistical Analysis 1: Comparison: Investigational vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 1.0, Bayesian logistic model — The posterior probably of non-inferiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 0.019, 95% CI 2-sided [-0.018 to 0.058] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Investigational vs Control; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.845, Bayesian logistic model — The posterior probably of superiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Success Rate of SF-36 PCS
Description: Success rate of SF-36 Health Survey include two components: the success rate of a physical component summary (PCS) and the success rate of a mental component summary (MCS). The success of SF-36 PCS was defined as: Post Score - Pre Score >= 0. The Success rate of SF-36 PCS is reported as the percentage of the participants who were classified as a success for SF-36 PCS.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable SF-36 PCS success status at 24 months, which leads to 264 subjects in the investigational group and 216 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 264 | 216
percentage of participants | 83.7 | 86.1
Statistical Analysis 1: Comparison: Investigational vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 0.936, Bayesian logistic model — The posterior probably of non-inferiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -0.047, 95% CI 2-sided [-0.113 to 0.021] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Success Rate of SF-36 MCS
Description: Success rate of SF-36 Health Survey include two components: the success rate of a physical component summary (PCS) and the success rate of a mental component summary (MCS). The success of SF-36 MCS were defined as: Post Score - Pre Score >= 0. The Success rate of SF-36 MCS is reported as the percentage of the participants who were classified as a success for SF-36 MCS.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable SF-36 MCS success status at 24 months, which leads to 264 subjects in the investigational group and 216 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 264 | 216
percentage of participants | 77.7 | 69.4
Statistical Analysis 1: Comparison: Investigational vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.1; p = 1.0, Bayesian logistic model — The posterior probably of non-inferiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 0.105, 95% CI 2-sided [0.020 to 0.190] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Investigational vs Control; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.992, Bayesian logistic model — The posterior probably of superiority was calculated and presented instead of the p-value; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Gait Success Rate
Description: Patient's gait was assessed by using Nurick's classification, and indicated either as normal or graded on a scale of 0 to 5. Success was defined as maintenance or improvement in the postoperative status as compared to the preoperative condition: Preoperative Score - Postoperative Score >= 0. The gait success rate is reported as the percentage of participants who had gait success.
Time Frame: 24 months
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable gait success status at 24 months, which leads to 270 subjects in the investigational group and 220 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 270 | 220
percentage of participants | 99.3 | 99.5

10. Secondary Outcome: Operative Time
Description: Operative time was recorded from skin incision to wound closure.
Time Frame: Time of operation, approximately 1.5 hrs.
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable information for operative time, which leads to 280 subjects in the investigational group and 265 subjects in the control group.
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Investigational | Control
Number analyzed (Participants) | 280 | 265
hrs | 1.5 (0.6) | 1.4 (0.5)
Statistical Analysis 1: Comparison: Investigational vs Control; Superiority comparison of the operative time in two treatment groups was assessed; Test type: Superiority or Other; p = 0.013, Bayesian logistic model — The posterior probably of superiority was calculated and presented instead of the p-value

11. Secondary Outcome: Blood Loss
Time Frame: During the time of operation, approximately 1.5 hours.
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable information for blood loss, which leads to 278 subjects in the investigational group and 263 subjects in the control group.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Investigational | Control
Number analyzed (Participants) | 278 | 263
ml | 50.5 (73.5) | 57.5 (68.1)
Statistical Analysis 1: Comparison: Investigational vs Control; Superiority comparison of the blood loss in two treatment groups was assessed; Test type: Superiority or Other; p = 0.769, Bayesian logistic model — The posterior probably of superiority was calculated and presented instead of the p-value

12. Secondary Outcome: Hospital Stay
Time Frame: During the time of hospital stay, average of 1 day.
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable information for hospital stay, which leads to 280 subjects in the investigational group and 265 subjects in the control group.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Investigational | Control
Number analyzed (Participants) | 280 | 265
days | 1.0 (0.5) | 1.0 (0.5)
Statistical Analysis 1: Comparison: Investigational vs Control; Superiority comparison of the hospital stay in two treatment groups was assessed; Test type: Superiority or Other; p = 0.273, Bayesian logistic model — The posterior probably of superiority was calculated and presented instead of the p-value

13. Secondary Outcome: Rate of Secondary Surgery at Index Level
Description: Secondary surgical procedures at the index level included revisions, removals, supplemental fixations and reoperations. Rate of secondary surgery at index level is reported as percentage of patients who had secondary surgeries at index level.
Time Frame: 24 months post-operation
Population: For this endpoint, the analysis consists of all subjects in the primary analysis dataset with 280 subjects in the investigational control and 265 subjects in the control group.
Measure: Number; unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 280 | 265
percentage of participants | 5.0 | 7.9

14. Secondary Outcome: Change of Neck Disability Index Score From Baseline
Description: The self-administered Neck Disability Index (NDI) Questionnaire was used to assess patient neck pain and ability to function. The NDI scale ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability). Change of NDI was defined as NDI at 24 month minus NDI at baseline.
Time Frame: Baseline and 24 months post-operation
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable NDI score at both baseline and 24 months, which leads to 270 subjects in the investigational group and 219 subjects in the control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Investigational | Control
Number analyzed (Participants) | 270 | 219
units on a scale
  NDI at baseline (n=280, 264) | 55.5 (14.7) | 56.4 (15.9)
  NDI at 24 months (n=270, 220) | 15.6 (18.3) | 22.4 (21.5)
  NDI change (n=270, 219) | -39.7 (21.0) | -33.9 (21.8)

15. Secondary Outcome: Change of Neck Pain Score From Baseline
Description: Numerical rating scales were used to evaluate neck pain intensity and frequency. Patients rated their neck pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be." Similarly, patients recorded their neck pain frequency on a scale from 0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time." The total neck pain score (0 to100) was the product of pain intensity and frequency scores. Change of neck pain score was defined as neck pain score at 24 months minus neck pain score at baseline.
Time Frame: Baseline and 24 months post-operation
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable neck pain score at both baseline and 24 months, which leads to 270 subjects in the investigational group and 219 subjects in the control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Investigational | Control
Number analyzed (Participants) | 270 | 219
units on a scale
  Neck Pain at baseline (n=280, 264) | 67.0 (20.8) | 69.3 (21.5)
  Neck Pain at 24 months (n=270, 220) | 10.6 (19.2) | 16.6 (24.4)
  Neck Pain Change (n=270, 219) | -56.6 (28.2) | -52.1 (28.3)

16. Secondary Outcome: Change of Arm Pain Score From Baseline
Description: Numerical rating scales were also used to evaluate arm pain intensity and frequency. Patients rated their arm pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be." Similarly, patients recorded their arm pain frequency on a scale from 0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time." The total arm pain score (0 to 100) was the product of pain intensity and frequency scores. Change of arm pain score was defined as arm pain score at 24 months minus arm pain score at baseline.
Time Frame: Baseline and 24 months post-operation
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable arm pain score at both baseline and 24 months, which leads to 268 subjects in the investigational group and 219 subjects in the control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Investigational | Control
Number analyzed (Participants) | 268 | 219
units on a scale
  Arm pain score at baseline (n=280, 264) | 59.6 (26.3) | 62.4 (28.5)
  Arm pain score at 24 months (n=268, 220) | 8.5 (18.3) | 14.2 (24.3)
  Arm pain score change (n=268, 219) | -52.0 (31.4) | -48.0 (32.7)

17. Secondary Outcome: Change of General Health Status -- SF-36 PCS From Baseline
Description: The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) was used to assess general health status. The SF-36 results were summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for PCS was between 0 and 100, with higher scores denoting better quality of life. Change of SF-36 PCS score was defined as PCS score at 24 months minus PCS score at baseline.
Time Frame: Baseline and 24 months post-operation
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable PCS score at both baseline and 24 months, which leads to 264 subjects in the investigational group and 216 subjects in the control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Investigational | Control
Number analyzed (Participants) | 264 | 216
units on a scale
  SF-36 PCS at baseline (n=279, 263) | 32.2 (7.4) | 32.0 (7.5)
  SF-36 PCS at 24 months (n=265, 218) | 46.6 (11.4) | 44.4 (12.0)
  SF-36 PCS change (n=264, 216) | 14.3 (11.6) | 11.9 (10.9)

18. Secondary Outcome: Change of General Health Status -- SF-36 MCS From Baseline
Description: The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) was used to assess general health status. The SF-36 results were summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for MCS was between 0 and 100, with higher scores denoting better quality of life. Change of SF-36 MCS score was defined as MCS score at 24 months minus MCS score at baseline.
Time Frame: Baseline and 24 months post-operation
Population: For this endpoint, the analysis consists of subjects in the primary analysis dataset with evaluable MCS score at both baseline and 24 months, which leads to 264 subjects in the investigational group and 216 subjects in the control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Investigational | Control
Number analyzed (Participants) | 264 | 216
units on a scale
  SF-36 MCS at baseline (n=279, 263) | 44.5 (11.5) | 42.7 (12.4)
  SF-36 MCS at 24 months (n=265, 218) | 52.6 (9.6) | 50.2 (11.1)
  SF-36 MCS change (n=264, 216) | 8.1 (12.3) | 7.2 (13.9)

ADVERSE EVENTS:
Time Frame: up to 24 months
Description: The adverse events, originally collected in FDA proposed categories, were grouped into organ systems.
Arm/Group | Investigational | Control
Serious Adverse Events (participants affected / at risk) | 133/280 | 98/265
Other Adverse Events (participants affected / at risk) | 242/280 | 211/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational (N=280) | Control (N=265)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 2 (2)
Cardiac Disorders (Cardiac disorders) | 9 (10) | 7 (8)
Dysphagia/Dysphonia (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 13 (22) | 12 (20)
Infection (Infections and infestations) | 11 (17) | 8 (8)
Neurological (Nervous system disorders) | 35 (52) | 27 (32)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 1 (1)
Trauma (Injury, poisoning and procedural complications) | 20 (22) | 10 (10)
Urogenital (Renal and urinary disorders) | 15 (20) | 4 (4)
Vascular (Vascular disorders) | 6 (7) | 0 (0)
Wound (Non-Infectious) (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Dysphagia/Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Heterotopic Ossification (Musculoskeletal and connective tissue disorders) | 11 (13) | 8 (12)
Implant Events (General disorders) | 4 (4) | 0 (0)
Neck and/or Arm Pain (Musculoskeletal and connective tissue disorders) | 37 (52) | 24 (36)
Non-Union (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)
Spinal Events (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Spinal Events (Musculoskeletal and connective tissue disorders) | 40 (77) | 31 (54)
Spinal Events (Nervous system disorders) | 1 (1) | 2 (3)
Other (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Other (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Other (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Other (Eye disorders) | 3 (5) | 1 (1)
Other (General disorders) | 1 (1) | 2 (2)
Other (Immune system disorders) | 1 (1) | 3 (3)
Other (Injury, poisoning and procedural complications) | 9 (9) | 3 (3)
Other (Investigations) | 3 (5) | 1 (2)
Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Other (Nervous system disorders) | 3 (3) | 2 (3)
Other (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Other (Psychiatric disorders) | 6 (8) | 5 (6)
Other (Surgical and medical procedures) | 3 (4) | 2 (2)
Other (Vascular disorders) | 1 (1) | 0 (0)
Other Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Other Pain (Eye disorders) | 1 (1) | 0 (0)
Other Pain (General disorders) | 3 (3) | 3 (4)
Other Pain (Injury, poisoning and procedural complications) | 10 (11) | 6 (7)
Other Pain (Musculoskeletal and connective tissue disorders) | 27 (38) | 16 (21)
Other Pain (Nervous system disorders) | 10 (12) | 2 (2)
Other Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational (N=280) | Control (N=265)
Anatomical/technical difficulty (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac Disorders (Cardiac disorders) | 8 (11) | 11 (12)
Dysphagia/Dysphonia (Gastrointestinal disorders) | 19 (21) | 21 (22)
Dysphagia/Dysphonia (Nervous system disorders) | 1 (1) | 0 (0)
Dysphagia/Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 25 (33) | 30 (48)
Heterotopic Ossification (Musculoskeletal and connective tissue disorders) | 16 (18) | 7 (9)
Implant Events (General disorders) | 12 (13) | 5 (5)
Infection (Infections and infestations) | 28 (40) | 22 (29)
Neck and/or Arm Pain (Musculoskeletal and connective tissue disorders) | 125 (223) | 113 (177)
Neurological (Nervous system disorders) | 116 (190) | 92 (185)
Non-Union (Musculoskeletal and connective tissue disorders) | 0 (0) | 24 (24)
Other (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Other (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Other (Ear and labyrinth disorders) | 5 (6) | 1 (2)
Other (Endocrine disorders) | 2 (3) | 2 (2)
Other (Eye disorders) | 3 (3) | 2 (2)
Other (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other (General disorders) | 11 (12) | 11 (14)
Other (Immune system disorders) | 6 (7) | 1 (1)
Other (Infections and infestations) | 0 (0) | 1 (1)
Other (Injury, poisoning and procedural complications) | 13 (14) | 4 (4)
Other (Investigations) | 15 (16) | 6 (7)
Other (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Other (Musculoskeletal and connective tissue disorders) | 17 (19) | 8 (9)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Other (Nervous system disorders) | 5 (6) | 12 (14)
Other (Psychiatric disorders) | 17 (21) | 16 (23)
Other (Renal and urinary disorders) | 0 (0) | 1 (1)
Other (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Other (Skin and subcutaneous tissue disorders) | 12 (13) | 10 (11)
Other (Social circumstances) | 2 (2) | 0 (0)
Other (Surgical and medical procedures) | 1 (1) | 2 (2)
Other (Vascular disorders) | 1 (1) | 0 (0)
Other Pain (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Other Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Other Pain (Eye disorders) | 1 (1) | 1 (1)
Other Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Other Pain (General disorders) | 6 (6) | 13 (13)
Other Pain (Injury, poisoning and procedural complications) | 17 (23) | 16 (20)
Other Pain (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Other Pain (Musculoskeletal and connective tissue disorders) | 88 (121) | 80 (122)
Other Pain (Nervous system disorders) | 43 (50) | 32 (35)
Other Pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Other Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 16 (22)
Spinal Events (Musculoskeletal and connective tissue disorders) | 50 (91) | 27 (42)
Spinal Events (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal Events (Nervous system disorders) | 1 (1) | 1 (1)
Trauma (Injury, poisoning and procedural complications) | 44 (49) | 30 (34)
Urogenital (Renal and urinary disorders) | 16 (22) | 6 (7)
Vascular (Vascular disorders) | 6 (6) | 4 (4)
Wound(Non-Infectious) (Injury, poisoning and procedural complications) | 20 (29) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less